CLINICAL TRIAL: NCT03994198
Title: Monitoring Exercise Performance and Mitigating Training Stress in Endurance-trained Cyclists
Brief Title: Effect of Protein Quality During Overreaching in Trained Cyclists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Stuart Phillips, Professor, McMaster University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: HIREB 3036
Record Dates: First submitted 2019-06-19; First posted 2019-06-21 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Muscle Protein Synthesis
MeSH Terms: interventions — Lactalbumin

STUDY DESIGN:
Intervention Model Description: Randomized cross-over design
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants and the investigators will be blinded the the supplement type, only the LPI will have the codes to decipher the supplement type. Supplements are referred to as A and B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alpha-lactalbumin (Experimental): Participants will consume 60 g of alphalactalbumin (fraction of whey protein) for 3 training days.
  Interventions: Dietary Supplement: Alpha-lactalbumin
- Collagen peptides (Active Comparator): Participants will consume 60 g of collagen peptides for 3 training days.
  Interventions: Dietary Supplement: Collagen peptides

INTERVENTIONS:
Dietary Supplement: Alpha-lactalbumin — A protein fraction of whey protein, higher in tryptophan
  Arms: Alpha-lactalbumin
Dietary Supplement: Collagen peptides — Collagen peptides from bovine sources
  Arms: Collagen peptides

SUMMARY:
Athletes frequently undertake periods of intensified training commonly referred to as "overreaching." These training periods acutely decrease performance, with the expectation that performance will rebound and improve after a short recovery. Yet, overreaching does not always improve performance and may be a precursor to overtraining syndrome, a long-term decrement in performance. A nutritional intervention focused on the adoption of 'best practices' for protein feeding (optimal timing, dose, and quality) could help reduce the stress of overreaching, reduce the likelihood of developing overtraining syndrome, and augment adaptations to intensified exercise. While the nutrition study is our main interest, the investigators first want to validate the measurement of exercise performance. Accordingly, this project consists of two related studies: (1) the assessment of short time trials for reliability and validity; and (2) the assessment of optimal protein feeding to decrease the stress of overreaching and improve outcomes following training.

DETAILED DESCRIPTION:
Endurance-trained athletes frequently undergo periods of overreaching (increased training loads) to improve performance. In study 1, the investigators will determine whether 4-min and 20-min time trials are repeatable and whether they (individually or collectively) relate to 1-hour time trial performance. For Study 2, the investigators propose that proper nutrition (with a focus on the dose, timing, and quality of protein) can help mitigate the stress of overreaching, which will improve performance. Thus, the investigators will compare the effects of two diets that differ in terms of protein servings (dose, timing, quality). In Study 2, skeletal muscle biopsies will be collected to determine how dietary protein intervention impacts the quality and quantity of skeletal muscle mitochondria in response to intense training.

For study 1, the objective is to determine the reliability and validity of 4-min and 20-min time trial performance (mean power output).

For study 2, the objective is to (1) determine whether following an optimal protein diet during a period of intense training will, relative to a typical diet: (1) improve measures of exercise performance, (2) improve sleep quality, psychological wellbeing, and immune function, (3) improve the quality and quantity of skeletal muscle mitochondria.

Study 1 is a reliability and validity experiment designed to assess the key outcome measure in study 2.

Study 2 is a randomized, crossover study. Participants will, in a randomized order, complete both conditions, separated by a 4-day washout period.

ELIGIBILITY:
Inclusion Criteria:

* non-smokers
* non-diabetic
* Participants had to be training regularly (performing aerobic exercise at least 4 times per week, including regular cycling exercise)
* Generally healthy

Exclusion Criteria:

* consuming excessive alcohol (>21 units per week)
* use of an investigational drug or nutraceutical in the previous 30 days
* dairy allergy
* history of significant loss or gain of body mass in the past 6 months (>2kg)
* regular use of non-steroidal anti-inflammatory drugs
* infectious disease, and/or the presence of any relevant disease (e.g., gastrointestinal, cardiovascular, neuromuscular, etc.).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Rate of myofibrillar muscle protein synthesis | 12 days
  Rate of myofibrillar and protein synthesis (%/day)
Rate of Sarcoplasmic muscle protein synthesis | 12 days
  Rate of sarcoplasmic muscle protein synthesis (%/day)

SECONDARY OUTCOMES:
Plasma amino acids | 1 x 1 hour
  Measurement of plasma amino acids 1 hour following ingestion of each beverage
Sleep efficiency (%) | 12 days
  Measured by Actigraphy
Sleep fragmentation | 12 days
  Measured by Actigraphy
Wake after sleep onset (WASO) in minutes | 12 days
  Measured by Actigraphy
Total sleep time (min) | 12 days
  Measured by Actigraphy

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Phillips, PhD, Principal Investigator — McMaster University
Locations (1):
- Ivor Wynne Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No